CLINICAL TRIAL: NCT02847104
Title: Impact of a Paper-based Dynamic Insulin Infusion Protocol on Glycemic Variability, Time in Target and Hypoglycemic Risk: a Stepped Wedge Trial in Medical ICU Patients
Brief Title: Medical ICU Paper-based Dynamic Insulin Protocol
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: VARIREA
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Stress Hyperglycemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- dynamic insulin protocol: patients received intravenous insulin infusion according to a dynamic insulin protocol
  Interventions: Other: dynamic insulin protocol
- static insulin protocol: patients received intravenous insulin infusion according to a static insulin protocol
  Interventions: Other: static insulin protocol

INTERVENTIONS:
Other: dynamic insulin protocol — Adaptation of insulin infusion rate according to hourly capillary blood glucose and dynamic insulin protocol
  Groups: dynamic insulin protocol
Other: static insulin protocol — Adaptation of insulin infusion rate according to hourly capillary blood glucose and static insulin protocol
  Groups: static insulin protocol

SUMMARY:
Intensive care unit (ICU) patients commonly display hyperglycemia, even without previously known diabetes. It was demonstrated that hyperglycemia was associated with increased hospital mortality in various medical and surgical ICU situations. However, discrepant results from recent randomized, clinical trials of tight blood glucose control in ICUs have not allowed conclusions regarding whether there is a causal link between hyperglycemia and ICU mortality. In addition to the mean blood glucose level, glucose variability has recently been emphasized as an independent predictor of ICU and hospital mortality. This concept has been described in a wide variety of medical, surgical and trauma ICU patients. In all of these settings, glycemic variability was measured with various indices but was steadily associated with ICU and/or hospital mortality in non-diabetic ICU patients. Conversely, glycemic variability was either weakly or not associated with mortality in ICU patients with previously known diabetes. Notably, all of these data have been observational, and interventional trials remain lacking to assess the impact of glycemic variability reduction on ICU mortality and thus to demonstrate causality. However, glycemic variability was considered sufficiently important to be mentioned in recent international guidelines for the management of hyperglycemia in critically ill patients. In these publications, experts from the American College of Critical Care Medicine emphasized that glycemia should be maintained at less than 9.9 mmol/L in ICU patients while avoiding hypoglycemia and minimizing glycemic variability. To achieve these goals, computer-based insulin infusion protocols have demonstrated their superiority to paper-based protocols. Glucose concentrations, variation per unit of time between the last and current glucose measurements, insulin dosage, and carbohydrate intake were the main input variables used in these different computerized algorithms. However, such protocols are not widely available because commercial systems have licensing fees and academic protocols do not always go beyond the pilot phase.

To address this issue, the investigators adapted a previously validated, paper-based, dynamic protocol (DP) to an actual recommended glycemic target range. Our aim was to assess the efficacy, safety, feasibility and acceptance by nurses of this dynamic insulin protocol, compared to a paper-based, sliding scale static protocol (SP).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patient admitted to intensive care unit
* Intensive care unit stay > 48 hours
* Stress hyperglycemia above 9.9 mmil/L indicating the need of continuous intravenous insulin infusion

Exclusion Criteria:

* Previous diabetes
* Acute metabolic event (ketoacidosis or hyperosmolarity)
* Insulin/dextrose infusion for hyperkalemia treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective trial involved adult patients who were admitted to the medical intensive care department of a French university hospital to compare the effects of two continuous intravenous insulin infusion (CIII) protocols on glycemic variability. According to the local protocol, patients with two consecutive capillary blood glucose measurements greater than 180 mg/dL (9.9 mmol/L), one hour apart, were considered to require CIII and were included in the trial. All of the patients or their family members received written information about the trial.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
MAGE (mean amplitude of glycemic excursion) index | calculated during the 5 first days after beginning of insulin infusion

SECONDARY OUTCOMES:
MAG: mean absolute glucose change | calculated during the 5 first days after beginning of insulin infusion
LI: lability index | calculated during the 5 first days after beginning of insulin infusion
SD: standard deviation of glycemia | calculated during the 5 first days after beginning of insulin infusion
CV: coefficient of variation of glycemia | calculated during the 5 first days after beginning of insulin infusion
LBGI: low blood glucose index | calculated during the 5 first days after beginning of insulin infusion
HBGI: high blood glucose index | calculated during the 5 first days after beginning of insulin infusion
GRADE: glycemic risk assessment diabetes equation | calculated during the 5 first days after beginning of insulin infusion
M-Value | calculated during the 5 first days after beginning of insulin infusion
mean blood glucose | calculated during the 5 first days after beginning of insulin infusion
time spent in the target range (140 to 180 mg/dL - 7.7 to 9.9 mmol/L) | calculated during the 5 first days after beginning of insulin infusion
low blood glucose episodes (less than 80 and 60 mg/dL - 4.4 and 3.3 mmol/L) (n/patient) | measured during the 5 first days after beginning of insulin infusion
severe hypoglycemia (less than 40 mg/dL - 2.2 mmol/L) (n/patient) | measured during the 5 first days after beginning of insulin infusion
time before the first glucose value in the target range (h) | calculated during the 5 first days after beginning of insulin infusion

CONTACTS AND LOCATIONS:
Overall Officials: damien du cheyron, PhD, Study Chair — University Hospital, Caen

IPD SHARING:
Plan to Share IPD: Undecided